CLINICAL TRIAL: NCT00114686
Title: A Multicenter, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind, Phase III Study to Compare the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL®) Versus Placebo as Adjunct Therapy With Mood Stabilizers (Lithium or Divalproex) for the Treatment of Alcohol Dependence in Patients With Bipolar I Disorder
Brief Title: Efficacy and Safety of Quetiapine Fumarate (SEROQUEL®) in the Treatment of Alcohol Dependency in Patients With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D144AL00002
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar I Disorder; Alcohol Dependence
Keywords: Bipolar I Disorder; Alcohol Dependency
MeSH Terms: conditions — Alcoholism | interventions — Quetiapine Fumarate; Lithium; Valproic Acid

INTERVENTIONS:
Drug: Quetiapine fumarate
Drug: lithium
Drug: divalproex

SUMMARY:
The purpose of this study is to determine whether treatment with Quetiapine Fumarate (SEROQUEL) in conjunction with mood stabilizers (Lithium or Divalproex) for 12 weeks helps patients who have Bipolar I Disorder with Alcohol Dependence

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Bipolar I Disorder with Alcohol dependence
* Outpatient Status
* Recent history of heavy drinking

Exclusion Criteria:

* Unstable medical illness
* Recent antipsychotic use
* Poorly controlled Diabetes Mellitus or Diabetes related illness

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of heavy drinking days from Baseline to Week 12, as derived from the Timeline Followback (TLFB) scale

SECONDARY OUTCOMES:
Change in the mean number of standardized drinks per day from Baseline to Week 12 & to monthly intervals, as derived from the TLFB scale
Change in manic symptoms as assessed by the change from Baseline to each visit in the Young Mania Rating Scale (YMRS) total score

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (38):
- United States (38):
  - Research Site, Cerritos, California
  - Research Site, San Diego, California
  - Research Site, New Haven, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Orlando, Florida
  - Research Site, Eagle, Idaho
  - Research Site, Shreveport, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Moorestown, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Research Triangle Park, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Media, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin